CLINICAL TRIAL: NCT00933309
Title: The Impact of Obesity and Obesity Treatments on Breast Cancer: A Phase I Trial of Exemestane With Metformin and Rosiglitazone for Postmenopausal Obese Women With ER+ Metastatic Breast Cancer
Brief Title: The Impact of Obesity and Obesity Treatments on Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0284
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast; Obese; Obesity Treatment; Exemestane; Aromasin; Metformin and Rosiglitazone; Avandamet; Postmenopausal; Hormone-sensitive; Hormone-receptive-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — exemestane; rosiglitazone-metformin combination; Metformin; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Exemestane alone
  Interventions: Drug: Exemestane
- Group 2 (Experimental): Exemestane plus Avandamet
  Interventions: Drug: Exemestane; Drug: Avandamet

INTERVENTIONS:
Drug: Exemestane — 25 mg tablets orally once a day
  Other Names: Aromasin®
Drug: Avandamet — Beginning dose 2 mg rosiglitazone with 500 mg metformin hydrochloride (2mg/500 mg) tablets taken orally once a day
  Other Names: Metformin plus rosiglitazone; Rosiglitazone and Metformin
  Arms: Group 2

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Avandamet that can be given in combination with exemestane to patients who are obese and postmenopausal with hormone-receptive-positive breast cancer that has spread to other parts of the body.

DETAILED DESCRIPTION:
The Study Drugs:

Exemestane decreases the ability of estrogen to help cancer cells grow. This could cause the cancer cells to die.

Avandamet contains two drugs commonly used to control blood sugar levels in patients with diabetes (metformin and rosiglitazone).

If you are found to be eligible to take part in this study, the dose of Avandamet you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of Avandamet. Each new group will receive a higher dose of Avandamet than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of Avandamet is found.

All participants will receive the same dose level of exemestane.

Study Drug Administration:

The study drug(s) will be given in 28-day "cycles."

You will take an exemestane tablet by mouth every day. You will also take tablets of Avandamet by mouth 1 or 2 times a day depending on the dose level to which you are assigned. You should take Avandamet at meals.

Study Visits:

On Day 1 of Cycles 2, 3, and 4, and then every 3 months after that, the following tests and procedures will be performed:

* You will have a physical exam, including a measurement of your weight and vital signs.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you may have taken or may be taking.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests. This blood draw can be done up to 3 days before each cycle.
* Blood (about 1 teaspoons) will be drawn for blood sugar tests. If you have a history of diabetes, you will need to fast for 8 hours before these blood sugar tests.

Every 3 months, you will have scans to check the status of the disease. The scan performed will depend on where the disease is located in the body.

Every 3 months, you will also have an echocardiogram (ECHO) or a multi-gated acquisition (MUGA) scan to test your heart function.

Additional Blood Draws:

Blood (about 1 teaspoon each time) will also be drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug(s) in the body at different time points. Blood will be drawn for PK testing before you take the study drug(s) and 1, 3, 6, 12, and 23 hours after you take the study drug(s) on Days 1, 8, and 15 of Cycle 1.

Length of Study:

You may take the study drug(s) for as long as the disease is stable and/or responding. You may be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Exemestane and Avandamet are FDA approved and commercially available. Exemestane is approved for the treatment of metastatic breast cancer. Avandamet is approved for the treatment of diabetes. The use of this drug combination is investigational.

Up to 24 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight or obese postmenopausal women with a history of biopsy-proven estrogen receptor positive and/or progesterone receptor positive breast cancer and clinical evidence of metastatic disease. Overweight and obesity are defined by the WHO as a BMI of 25 - 29.9 and >/= 30 kg/m^2 respectively. Postmenopausal status is defined by one of the following: a) no spontaneous menses for over 1 year, in women >55 years; Continued in inclusion criterion # 2.
2. Continuation from inclusion #1: b) no spontaneous menses within the past 1 year in women </= 55 years with postmenopausal gonadotrophin levels (LH and FSH levels > 40 IU/L) or postmenopausal estradiol levels (<10 pg/mL); or c) bilateral oophorectomy.
3. Prior endocrine therapy, biologic therapy and chemotherapy are allowed, either in the adjuvant setting or for metastatic breast cancer.
4. Prior exemestane, metformin, or rosiglitazone is allowed if taken longer than 7 days prior to enrollment.
5. Localized radiotherapy, which does not influence the signal of evaluable lesion, is allowed prior to the initiation of study medications.
6. Performance status </= 2 ECOG.
7. Absolute neutrophil count (ANC) >/= 1000/µl, platelets >/= 75,000/µl, hemoglobin >/= 8.5 gm/dL; serum creatinine < 1.4 mg/dL; bilirubin < 1.8 mg/dL; ALT or AST </= 2.5 x ULN if no demonstrable liver metastases or </= 5 x ULN in presence of liver metastases; alkaline phosphatase < 3 x upper limit of normal; calcium </= 11.0 mg/dL.
8. Patients must be competent to give informed consent and to state that they understand the investigational nature of the proposed treatment.

Exclusion Criteria:

1. Extensive radiotherapy within previous 4 weeks (greater than or equal to 30% of marrow-bearing bone, e.g., whole pelvis or half spine).
2. Uncontrolled diabetes mellitus (hemoglobin A1C > 9 or random plasma glucose > 400 mg/dL).
3. History of acromegaly, Cushing's syndrome, Cushing's disease, Addison's disease (treated or untreated).
4. Patients with unstable angina, uncontrolled ischemic cardiac disease or symptomatic congestive heart failure (e.g. Class III or IV New York Heart Association's Functional Classification).
5. Concurrently receiving and are unwilling to discontinue hormonal (estrogen with or without progesterone) replacement therapy.
6. Other investigational drugs within the past 3 weeks or concurrently.
7. Patients with known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Laboratory results sustained at: International normalized ratio (INR) > 1.6; ALT or AST > 2.5 x ULN if no demonstrable liver metastases or > 5 x ULN in presence of liver metastasis; No more than 3 retests within screening period
9. Patients with known diagnosis of human immunodeficiency virus (HIV) infection.
10. Patients who received chemotherapy within 3 weeks (6 weeks for nitrosourea or mitomycin-C). Acute toxicities from prior therapy must have resolved to Grade </= 1 with the exception of fatigue, alopecia, or anemia.
11. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol e.g., severe renal or hepatic impairment or currently unstable or uncompensated respiratory or cardiac conditions.
12. History of hypersensitivity to active or inactive excipients of the study medications - exemestane or metformin.
13. Untreated or clinically unstable central nervous system involvement. A patient with adequately treated brain metastases would be eligible one month after completion of surgery and/or radiation therapy if she is clinically stable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Day 1 of each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Esteva, MD, PhD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org